CLINICAL TRIAL: NCT03038321
Title: Solifenacin vs Levofloxacin vs Lornoxicam for Management of Intravesical Instillation of Bacillus Calmette-Guerin (BCG) Side Effects A Single Blinded Randomised Controlled Study
Brief Title: Solifenacin, Levofloxacin or Lornoxicam, Which Is Ideal for Management of Intravesical Instillation BCG Side Effects?
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Abdelwahab Hashem, Urology Msc, Oncology fellow at Urology and Nephrology Center, Principal Investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R/17.01.02
Record Dates: First submitted 2017-01-15; First posted 2017-01-31 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-03

CONDITIONS: Non-Muscle-invasive Bladder Cancer (NMIBC); Bacillus Calmette-Guerin (BCG) Cystitis; Intra-vesical Instillation
Keywords: BCG Cystitis; Bladder Cancer; Levofloxacin; Solifenacin; Lornoxicam
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms; Cystitis; Urinary Bladder Neoplasms | interventions — Ofloxacin; lornoxicam

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- solifenacin (Active Comparator): (Sofenacin ''solifenacin 10 m'') [Marcyrl Pharmaceutical Industries - Egypt]
  Interventions: Drug: sofenacin
- levofloxacin (Active Comparator): (Tavanic ''levofloxacin 500 mg'') [Sanofi-Aventis - Egypt]
  Interventions: Drug: Tavanic
- lornoxicam (Active Comparator): (Xefo ''lornoxicam 8 mg'') [Multi-Apex - Egypt, under license of: NYCOMED, Austria]
  Interventions: Drug: Xefo

INTERVENTIONS:
Drug: sofenacin — solifenacin 10 mg, 6 hours after IVI of BCG and continue for another 2 days post instillation
  Other Names: Solfenacin 10 mg
  Arms: solifenacin
Drug: Tavanic — levofloxacin 500 mg, 6 hours after IVI of BCG and continue for another 2 days post instillation.
  Other Names: levofloxacin 500
  Arms: levofloxacin
Drug: Xefo — lornoxicam 8 mg, 6 hours after IVI of BCG and continue for another 2 days post instillation.
  Other Names: lornoxicam
  Arms: lornoxicam

SUMMARY:
Compare the different supposed clinical treatment of side effects associated with intravesical BCG by levofloxacin (quinolones) vs solifenacin (selective anti-muscarinic) vs lornoxicam (NSAID)

DETAILED DESCRIPTION:
For urothelial carcinoma (UC), which accounts for over 90% of bladder cancers, more than 70% of bladder cancer patients present with non-muscle-invasive disease. Approximately 40-80% of these tumors will recur within the first year, of which 10-25% will progress to muscle-invasive disease.

Intravesical treatments with cytotoxic chemotherapy and immunotherapy have become the mainstay following transurethral resection (TUR). Increasing knowledge of BCG use allows for effective management of these once debilitating side effects. The majority of patients will still experience cystitis-like symptoms to some degree, including urinary frequency (71%), cystitis (67%), fever (25%), and hematuria (23%).

Oxybutynin increases in fever, flu-like symptoms, dry mouth and constipation. However, in this study oxybutynin started the night before treatment causing an element of incomplete bladder emptying and allowing an increased BCG dwell time. We think that these effect can be reversed by use anticholinergic 6 hours post BCG instillation Anti-inflammatory drugs significantly reduced BCG-induced granulocyte activation and did not impair BCG-induced lymphocyte cytotoxicity against bladder tumor cells in mice. The committee of International Bladder Cancer Group (IBCG) recommend use of anti-inflammatory agents (NSAIDs) for treatment of non-bacterial or chemical cystitis and other systemic BCG side effect.

Fluoroquinolone with tuberculostatic properties, has been shown to significantly prolong survival in mice with BCG systemic infection and did not affect the antitumor efficacy of BCG. ofloxacin significantly decreased by 18.5% the incidence of class II or higher moderate and severe adverse events of BCG.

Because of sparse published studies on BCG side effect management, the 2016 European Association of Urology (EAU) guidelines management options for side effects associated with intravesical BCG modify the IBCG committee clinical practice without any degree of recommendation. So, in this study the investigators will try to fill the gap in the literature.

ELIGIBILITY:
Inclusion Criteria:

• Patients classified as intermediate or high risk of the bladder tumour

Exclusion Criteria:

* Patient over 80 years (natural decline in immune system function)
* Refuse to complete study requirements
* Contraindication to BCG therapy
* High post-void residual (PVR) above 85 ml
* American Urological Association (AUA) Symptoms score above 20
* Sensitivity to previously mentioned 3 drugs
* High serum creatinine

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Comparing the drugs efficacy on decreasing systemic and local side effects of BCG | 6 weeks
  __ Outcome Measure by Four-class classification grid of BCG adverse events

SECONDARY OUTCOMES:
Comparing the drugs effect on decreasing voiding and storage urinary symptoms of BCG | 6 weeks
  __ Outcome Measure by overactive bladder symptoms scores and American Urological Association Symptom Index
Prostatic specific antigen (PSA) change | 1 month and 3 months
  __ Outcome Measure by PSA measure 1 and 3 months post instillation
recurrence free survival | 1 year
  __ Outcome Measure by Number of patients surviving for one year without tumor recurrence will be counted and compared

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Abol-Enein, MD, Phd, Study Chair — Urology and Nephrology Center; Ahmed Mosbah, MD, Study Director — Urology and Nephrology Center; Ahmed Elhussein, MBBCH, Principal Investigator — Urology and Nephrology Center; Ahmed Elkarta, MBBCH, Principal Investigator — Urology and Nephrology Center; Mohamed Soltan, Principal Investigator — Urology and Nephrology Center
Locations (1):
- Urology and Nephrology Center, Al Mansurah, Aldakahlia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
meta-analyses by contact the Prof. Hassan Abol-Enein, MD, Phd (Study Chair)